CLINICAL TRIAL: NCT06287970
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Moderate to Severe Chronic Prostatitis/Chronic Pelvic Pain Syndrome (TASC-P Trial): a Randomized, Sham Controlled Trial.
Brief Title: TaVNS Improves the Symptoms of Patients With Moderate to Severe CP/CPPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiani Wu (Other)
Responsible Party: Sponsor-Investigator, Jiani Wu, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-250-KY
Record Dates: First submitted 2024-02-04; First posted 2024-03-01 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Prostatitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS Group (Experimental): Bilateral auricular points of Xin (CO15) and Shen (CO10) will be stimulated by electrical stimulation. A disperse-dense wave will be used with a frequency of 4Hz/20Hz, a pulse width of 0.2ms will be set, and the current intensity will be modulated by the tolerance of the patient.
  note: taVNS, transcutaneous auricular vagus nerve stimulation
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Sham-taVNS Group (Sham Comparator): Bilateral ear lobes will be stimulated by electrical stimulation. A disperse-dense wave will be used with a frequency of 4Hz/20Hz, a pulse width of 0.2ms and a current intensity of 0.1mA will be set.
  note: taVNS, transcutaneous auricular vagus nerve stimulation
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — In the experimental group, bilateral auricular point Xin (CO15) and auricular point Shen (CO10) will be stimulated, on where the vagus nerves distributed.
  Arms: taVNS Group
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation — In the control group, bilateral earlobes will be stimulated with no vagus nerve distribution.
  Arms: Sham-taVNS Group

SUMMARY:
This trial aims to evaluate the efficacy and safety of transcutaneous auricular vagus nerve stimulation (taVNS) for moderate to severe chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). This study is a prospective, randomized, controlled trial. A total of 68 patients with CP/CPPS will be recruited. After baseline assessment, the patients will be randomized into taVNS group (n = 34) and sham-taVNS group (n = 34). The intervention of two group will last for 4 weeks with a 8-week follow-up period after the treatment. The National Institutes of Health chronic Prostatitis Symptom Score index (NIH-CPSI), International Prostate Symptom Score Scale (IPSS), European quality of Life-5 Dimensions Questionnaire (EQ-5D), self-rating anxiety Scale (SAS) and self-rating depression scale (SDS) will be assessed. The adverse events during the whole study will be recorded detailedly.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with the diagnostic criteria of CP/CPPS of EAU or CAU, the clinical manifestations were recurrent and persistent prostate pain accompanied by abnormal urination and psychiatric symptoms, without infection or other obvious pathological conditions. The pain symptoms were mainly manifested as pain in the surrounding tissues centered on the prostate, and pain, swelling or discomfort in the scrotum, testis, lower abdomen, perineum, lumbosacral area, and medial thigh. Abnormal urination was characterized by frequent urination, urgent urination, urination pain, urethral burning, residual urination or white discharge from the urethra at the end of urination or defecation in the morning. The neuropsychiatric symptoms included dizziness and tinnitus, insomnia and dreams, anxiety and depression, and even impotence, premature ejaculation, and spermatorrhea. Symptoms lasting more than 3 months in the last six months
* 18 ≤ Age ≤ 50 years old
* NIH-CPSI ≥15 (patients with moderate to severe CP/CPPS)
* Signed informed consent and voluntarily participated in the trial

Exclusion Criteria:

* Patients with other diseases that cause urinary symptoms were excluded: Such as benign prostatic hyperplasia, testicular and epididymal and spermatic cord diseases, overactive bladder, neurogenic bladder, interstitial cystitis, glandular cystitis, sexually transmitted diseases, bladder tumors such as carcinoma in situ, prostate cancer, urinary male reproductive system tuberculosis, anorectal diseases, lumbar diseases, central and peripheral neuropathy, etc
* Patients with severe diseases of the heart, liver, kidney, hematopoietic system and poor nutritional status
* Patients with severe mental and emotional disorders, who were unable to cooperate with the study
* Patients who have been treated with CP/CPPS regimen in the past 4 weeks

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in National Institute of Health Chronic Prostatitis Symptom Index(NIH-CPSI) total score at week 4 | Baseline, week 4
  The NIH-CPSI scale scores range from 0 to 43, with higher scores indicating more severe symptoms. The NIH-CPSI total score will be recorded once a week during the treatment period.

SECONDARY OUTCOMES:
Change from baseline in National Institute of Health Chronic Prostatitis Symptom Index(NIH-CPSI) total score at week 8 and week 12 | Baseline, week 8 and 12
  The NIH-CPSI scale scores range from 0 to 43, with higher scores indicating more severe symptoms. The NIH-CPSI total score will be recorded once a week during the treatment and follow-up period
The changes from baseline of NIH-CPSI pain score, urinary score and quality of life score, respectively at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  The NIH-CPSI scores range from 0 to 43. The NIH-CPSI has three subscores: pain scores , urinary scores , and quality of life scores. The subscore of pain ranged from 0 to 21. The subscores of urination symptoms ranged from 0 to 10. The subscore of the effect of symptoms on quality of life ranges from 0 to 12. The higher the score, the more severe the symptoms. These subitem scores are specific to the symptoms of CP/CPPS and do not require other separate outcome measures. Each part of the NIH-CPSI score will be recorded weekly during the treatment and follow-up periods
Proportion of responders at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  Responder is defined as the patient with a decrease of ≥6 points in the NIH-CPSI total score compared with baseline. The proportion of responders will be calculated for each evaluation time point.
The change from baseline in International Prostate Symptom Score (IPSS) score at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  The IPSS scale scores range from 0 to 35, with higher scores indicating more severe symptoms. The total IPSS score will be recorded once a week during the treatment and follow-up period
The change from baseline in EuroQol Five Dimensions Questionnaire (EQ-5D) at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  The EQ-5D is mainly composed of two parts, the Descriptive System and the Visual Analogue Scale (VAS) . The description system of EQ-5D can generate a five-digit health status, which can be intuitively reflected in the five health dimensions. This health status can be converted into a single summary number (utility index value) according to the characteristics of the general population in a country/region, which can be used to reflect the health status. The Visual Analogue Scale (VAS) contains a vertical scale ranging from 0 to 100 to record the self-rated health status of the participants. The Visual Analogue Scale provides a quantitative description of respondents' perceptions of their overall health. The EQ-5D total score will be recorded once a week during the treatment and follow-up period
The change from baseline in Self-rating Anxiety Scale (SAS) at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  The standard score of the test result is obtained by summing the scores of the 20 items in the SAS scale, multiplying the resulting result by 1.25 and rounding to integer numbers. The cut-off value of the standard score is 53 points, with 53 to 62 points as mild depression, 63 to 72 points as moderate depression, and more than 73 points as severe depression. The total score of SAS will be recorded once a week during the treatment and follow-up period
The change from baseline in the Self-rating Depression Scale (SDS) at week 4, 8 and 12 | Baseline, week 4, 8 and 12
  The standard score of the test result is obtained by summing the scores of the 20 items in the SDS scale, multiplying the resulting result by 1.25 and rounding to integer numbers. The cut-off value of the standard score is 53 points, with 53 to 62 points as mild depression, 63 to 72 points as moderate depression, and more than 73 points as severe depression. The total score of SDS will be recorded once a week during the treatment and follow-up period

OTHER OUTCOMES:
Evaluation of patient expectations | Baseline before the randomization
  Patients will be asked before the randomization: ① Do you think transcutaneous vagal nerve stimulation will be effective? ② Do you think transcutaneous vagal nerve stimulation will help improve your symptoms of chronic prostatitis/chronic pelvic floor pain syndrome?
Blinding Evaluation | at the end of week 4
  Let the patient choose whether or not he or she has received the taVNS treatment after the treatment
Incidence of Treatment-Emergent Adverse Events | The 4-week treatment period
  Treatment-related adverse events will be recorded and evaluated between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospita, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article and any future publications from this study will be shared. This includes, but is not limited to: demographic information, clinical assessments, scores from the National Institutes of Health Chronic Prostatitis Symptom Score Index (NIH-CPSI), the International Prostate Symptom Score Scale (IPSS), the European Quality of Life Five-Dimensions Questionnaire (EQ-5D-5L), the Self-rating Anxiety Scale (SAS), and the Self-rating Depression Scale (SDS).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available starting 6 months after publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: De-identified data will be made available to qualified researchers upon reasonable request. Researchers must submit a methodologically sound research proposal to the corresponding author at jiani_wu@aliyun.com. Access to the data will be granted after the requester signs a formal data access agreement.